CLINICAL TRIAL: NCT04986631
Title: Pharmacokinetics and Pharmacodynamics of Topiramate for Weight Loss in Youth: PHARMATOP
Acronym: PHARMATOP
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEDS-2021-29920
Record Dates: First submitted 2021-07-16; First posted 2021-08-03 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Obesity, Childhood
MeSH Terms: conditions — Pediatric Obesity | interventions — Topiramate

STUDY DESIGN:
Intervention Model Description: Individuals in this pilot study will be 12-<18 years of age at enrollment. All participants will receive topiramate for 3.5 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Topiramate (Experimental): Individuals will receive 75 mg of topiramate daily. The dose will start at 25 mg daily for the first week. The second week participants will receive 50 mg daily. Starting at week 3 participants will take 75 mg daily.
  Interventions: Drug: Topiramate Tablets

INTERVENTIONS:
Drug: Topiramate Tablets — Topiramate intervention

SUMMARY:
Pediatric severe obesity is the fastest growing obesity category in the United States, and anti-obesity pharmacotherapies are promising adjuncts to lifestyle modification (LSM) for the treatment of this disease. While anti-obesity pharmacotherapies have overall been associated with mean weight loss, there is substantial variability in their individual-level effectiveness. While some patients lose a significant amount of weight with anti-obesity pharmacotherapies, others lose little or even gain weight.

Due to this well-recognized variability in individual-level response, the National Institutes of Health (NIH) has recognized the importance of using precision medicine approaches in order to optimize treatments for pediatric severe obesity. Pharmacometrics, which uses mathematical models to study medication dose-exposure (i.e. blood drug concentrations)-response relationships, is an emerging science that can help determine optimal dosing regimens based upon patient-specific characteristics. Pharmacometrics quantitates the interplay between pharmacokinetics (PK; drug dose-exposure associations) and pharmacodynamics (PD; drug exposure-response associations). Population PK (popPK), a type of PK, can be used to quantitate variability in drug exposure among individuals in order to help inform recommendations on therapeutic individualization (e.g. through tailored dosing). In this study, investigators will use popPK/PD modeling to characterize associations between anti-obesity pharmacotherapy dose, exposure, and changes in weight and weight-related outcomes in youth with severe obesity.

This study will focus on topiramate because this medication is commonly prescribed for weight loss in youth with severe obesity and has been associated with highly variable individual-level effectiveness.

DETAILED DESCRIPTION:
The weight loss achieved with topiramate occurs through several purported mechanisms including reductions in appetite, food cravings, and binge eating, and adverse alterations in taste for carbonated beverages. It is hypothesized that some of the individual-level effectiveness of this medication on weight loss response is secondary to patient-specific differences in these factors. In a 3.5-month pragmatic-based prospective cohort study (n=65), the investigators will develop a popPK model using sparse sampling by drawing a series of topiramate concentration measures over time in order to begin determining patient-specific factors that contribute to topiramate exposure variability. The investigators will also identity associations between topiramate exposure, changes in eating behaviors, and weight loss outcomes through PD models using regression techniques. It is hypothesized that patient-specific characteristics (i.e. age, body mass index (BMI), and sex) will explain some variability in topiramate exposure in youth, and that higher topiramate exposure will be associated with greater improvements in weight loss response and eating behaviors among youth prescribed this medicine for the treatment of pediatric severe obesity.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) </= 1.2 times the 95th percentile (age and sex-adjusted) and/or BMI >/= 35 kg/m2
* Ages 12 to < 18 years old
* Deemed appropriate candidates to receive topiramate (without contraindications) for weight loss by an obesity medicine specialist at the University of Minnesota

Exclusion Criteria:

* History of metabolic/bariatric surgery
* Obesity associated with a diagnosed genetic disorder (i.e. monogenic obesity, Prader-Willi, Bardet-Biedl syndrome)
* Clinically diagnosed hyperthyroidism or uncontrolled hypothyroidism as determined by local medical monitor (who is a board certified endocrinologist)
* History of acute angle closure glaucoma. Individuals with other types of glaucoma will need approval from the participant's ophthalmologist to be enrolled.
* History of nephrolithiasis
* History of seizures (aside from febrile seizures)
* Major psychiatric disorder as determined by local medical monitor
* History of bulimia nervosa or anorexia nervosa
* History of suicide attempt within the last year

  * History of active suicidal ideation or self-harm within the past 30 days
* Current or recent (< 6 months prior to enrollment) use of anti-obesity medication(s) defined as orlistat, phentermine, topiramate, combination phentermine/topiramate, liraglutide (or other glucagon-like peptide (GLP1-RA)), and/or combination naltrexone/bupropion (monotherapy use of naltrexone or bupropion is not an exclusion), unless participant has been on stable doses for >/= 6 months. Of note, if phentermine was increased from 15 mg daily to 18.75 mg daily during this period, it is not considered a dose increase.
* Current or recent (< 6 months prior to enrollment) use of medication(s) associated with weight gain (e.g. oral steroids, anti-psychotics), unless participant has been on stable doses of such medication(s) for ≥ 6 months
* Current or recent (< 6 months prior to enrollment) use of long-acting stimulant medications, unless participant has been on stable doses of such medication for ≥ 6 months. In terms of short-acting ADHD stimulant medications, the PI will determine eligibility based on weight and dose (no studies have shown this contributes to weight outcomes)
* Baseline bicarbonate < 18 mmol/L
* Baseline creatinine > 1.2 mg/dL
* Females: pregnant, planning to become pregnant, or, if sexually active, unwilling to use 2+ acceptable contraceptive methods during the study period

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 65 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2025-03-12 (Actual); Study Completion 2026-03-12 (Estimated)

PRIMARY OUTCOMES:
To determine associations between topiramate exposure and 3-month BMI change using pharmacodynamic modeling | 3 months
  Change in body mass index (BMI) as assessed by percent change in BMI from baseline to Month 3

CONTACTS AND LOCATIONS:
Overall Officials: Eric Bomberg, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Summary data that has been de-identified will be made available to other researchers
Supporting Information: Study Protocol, SAP, CSR

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-05-03): https://cdn.clinicaltrials.gov/large-docs/31/NCT04986631/Prot_SAP_002.pdf
  • Informed Consent Form (2023-06-13): https://cdn.clinicaltrials.gov/large-docs/31/NCT04986631/ICF_000.pdf